CLINICAL TRIAL: NCT06946511
Title: Exploratory Study of the Effects of Peptide PMS-001 on Long-Delay Recall in Patients With Moderate to Severe Dementia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, liu jun, Chief Physician, Director of the Department of Neurology, distinguished professor of the "Changjiang Scholars Program" of The Ministry of Education, doctoral supervisor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RuijinH-2025125
Record Dates: First submitted 2025-04-10; First posted 2025-04-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Dementia
Keywords: Dementia; Treatment
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PMS-001 Injection, 15mg (Experimental): Participants in this group will receive an injection of PMS-001 at a dose of 15mg. This group is designed to evaluate the efficacy and safety of PMS-001 at the lowest dose level.
  Interventions: Drug: Peptide PMS-001 Intravenous Injection
- PMS-001 Injection, 30mg (Experimental): Participants in this group will receive an injection of PMS-001 at a dose of 30mg. This group is designed to evaluate the efficacy and safety of PMS-001 at a moderate dose level.
  Interventions: Drug: Peptide PMS-001 Intravenous Injection
- PMS-001 Injection, 60mg (Experimental): Participants in this group will receive an injection of PMS-001 at a dose of 60mg. This group is designed to evaluate the efficacy and safety of PMS-001 at a higher dose level.
  Interventions: Drug: Peptide PMS-001 Intravenous Injection
- PMS-001 Injection, 75mg (Experimental): Participants in this group will receive an injection of PMS-001 at a dose of 75mg. This group is designed to evaluate the efficacy and safety of PMS-001 at the highest dose level.
  Interventions: Drug: Peptide PMS-001 Intravenous Injection
- Placebo (Placebo Comparator): Participants in this group will receive an injection of placebo. This group serves as a control to compare the effects of PMS-001 on long-delay recall and safety in patients with moderate to severe dementia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Peptide PMS-001 Intravenous Injection — Participants will receive intravenous injections of PMS-001.
  Arms: PMS-001 Injection, 15mg; PMS-001 Injection, 30mg; PMS-001 Injection, 60mg; PMS-001 Injection, 75mg
Drug: Placebo — The control group will receive a placebo, which is the blank excipient (mannitol) of the injectable PMS-001.
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled study. Patients will be randomly assigned to either the peptide intervention group (with dose escalation at 15mg, 30mg, 60mg, and 75mg) or the placebo control group. After learning and training, participants will receive an injection of PMS-001. The efficacy and safety of the intervention will be assessed at 1 hour, 1 day, 3 days, and 1 week post-intervention. This study aims to evaluate the effects of PMS-001 on improving long-delay recall in patients with moderate to severe dementia, as well as its safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged 60 to 80 years (inclusive) at the time of screening, regardless of gender.
2. Participants must have a Clinical Dementia Rating (CDR) total score > 1, indicating moderate to severe dementia.
3. Participants must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of other neurological diseases that may cause cognitive decline, such as cerebrovascular disease, encephalitis, brain tumors, traumatic brain injury, epilepsy, Parkinson's disease, etc.
2. Presence of metabolic diseases that may cause cognitive decline, such as anemia, thyroid dysfunction, folate and vitamin B12 deficiency, etc.
3. Presence of severe psychiatric disorders, such as major depression.
4. History of carbon monoxide poisoning.
5. Presence of acute or severe life-threatening diseases.
6. Presence of severe visual, auditory, or language impairments that would prevent the completion of neuropsychological assessments.
7. Current use of psychotropic medications or a history of substance abuse.
8. Individuals with specific allergy histories, or those with a history of allergies to two or more medications, foods (such as milk), or pollen (excluding untreated, asymptomatic seasonal allergies), or known allergies to components of the study drug or similar agents.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of Peptide PMS-001 in improving long-delay recall in patients with moderate to severe dementia. | Clinical assessments will be conducted at baseline, and then at 1 hour, 1 day, 3 days, and 1 week after administration of the intervention.
  The primary outcome will be specifically assessed using the sum of the long-delay recall scores from the following evaluation scales:
  The Auditory Verbal Learning Test - Huashan Version (AVLT-H): The long-delay recall score (AVL-LR) is the number of words correctly recalled after a 20-minute delay. The AVL-LR score ranges from 0 to 12, with higher scores indicating better memory performance and lower scores suggesting more significant memory impairment.
  Logical Memory Story A (LM-A) from the Wechsler Memory Scale - III (WMS-III): The long-delay recall score for LM-A measures the participant's ability to recall the story after a delay. The LM-A long-delay recall score ranges from 0 to 25, with higher scores indicating better memory function and lower scores pointing to memory deficits.
  The changes in participants' total scores, which are the sum of the long-delay recall scores from both AVLT-H and WMS-III LM-A, before and after treatment will be evaluated using these scales.

SECONDARY OUTCOMES:
Assessment of the impact of Peptide PMS-001 on overall cognitive function in patients with moderate to severe dementia | Clinical assessments will be conducted at baseline, and then at 1 hour, 1 day, 3 days, and 1 week after administration of the intervention.
  Evaluation Scales: Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point test that assesses multiple cognitive domains, including memory, attention, language, and visuospatial skills. The score ranges from 0 to 30, with higher scores indicating better cognitive function and lower scores suggesting worse cognitive outcomes.
Assessment of the impact of Peptide PMS-001 on executive function in patients with moderate to severe dementia. | Clinical assessments will be conducted at baseline, and then at 1 hour, 1 day, 3 days, and 1 week after administration of the intervention.
  Evaluation Scales: Trail Making Test B (TMT-B). The TMT-B is a widely used neuropsychological test that measures cognitive flexibility, attention, and processing speed. In this test, participants are required to connect a series of alternating numbers and letters as quickly as possible. The score is typically the time taken to complete the test, with a minimum possible score of 0 seconds (indicating no time taken, which is practically impossible) and no upper limit, as completion time can vary widely among individuals.
  A lower TMT-B score (shorter completion time) indicates better performance, reflecting higher cognitive flexibility, better attention, and faster processing speed.
  A higher TMT-B score (longer completion time) suggests more significant cognitive impairment, particularly in the areas of cognitive flexibility and attention.
Assessment of the impact of Peptide PMS-001 on language function in patients with moderate to severe dementia. | Clinical assessments will be conducted at baseline, and then at 1 hour, 1 day, 3 days, and 1 week after administration of the intervention.
  Evaluation Scales: Boston Naming Test (BNT). The BNT is a widely used neuropsychological test designed to assess language function, specifically the ability to name objects and concepts. It consists of a series of line drawings that participants are asked to name. The BNT typically includes 30 items, and the score ranges from 0 to 30, with each correctly named item contributing 1 point.
  A higher BNT score (closer to 30) indicates better language function and naming ability, suggesting that the participant has less difficulty with word retrieval and object naming.
  A lower BNT score (closer to 0) suggests more significant language impairment, which may be indicative of difficulties in word finding or naming, often seen in conditions such as aphasia or cognitive decline.
Assessment of the impact of Peptide PMS-001 on visuospatial function in patients with moderate to severe dementia. | Clinical assessments will be conducted at baseline, and then at 1 hour, 1 day, 3 days, and 1 week after administration of the intervention.
  Evaluation Scales: Clock Drawing Test (CDT). The CDT is a widely used neuropsychological test that assesses cognitive function, particularly executive function and visuospatial abilities. In this test, participants are asked to draw a clock, including all the numbers and setting the time to a specific hour (e.g., 10 past 11). The score ranges from 0 to 20, with higher scores indicating better cognitive function and visuospatial skills
Assessment of the impact of Peptide PMS-001 on event-related potentials in patients with moderate to severe dementia. | Clinical assessments will be conducted at baseline, and then at 1 hour, 1 day, 3 days, and 1 week after administration of the intervention.
  Evaluation Method: Event-Related Potentials (ERP). Event-Related Potentials (ERPs) are electrophysiological neural responses time-locked to specific stimuli and are widely used to assess various cognitive processes。 A larger amplitude generally indicates a stronger neural response to a stimulus. For example, in cognitive tasks, a larger P300 amplitude (a positive wave occurring around 300ms after a stimulus) is often associated with increased attention and cognitive processing。

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided